CLINICAL TRIAL: NCT06106191
Title: Integrative Mindfulness-Based Predictive Approach for Chronic Low Back Pain Treatment
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Worcester Polytechnic Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-44407; UG3NS135168 (NIH)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low-back Pain
Keywords: Mindfulness based stress reduction (MBSR); Machine learning (ML); Biopsychosocial data; PEG (Pain, Enjoyment, General activity); Pain interference; Pain intensity; Depression
MeSH Terms: conditions — Pain; Motor Activity; Depression | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness based stress reduction (MBSR) program (Experimental): Participants will be enrolled in a 8-week mindfulness clinical pain program + Primary Care Provider (PCP) Usual Care.
  Interventions: Behavioral: Mindfulness meditation; Other: Perspectives on pain; Other: Discussion

INTERVENTIONS:
Behavioral: Mindfulness meditation — Ordinary activities like breathing, eating, and walking are turned into a meditation by creating greater awareness of the moment-to-moment sensations, emotions, thoughts and behaviors that arise during these activities.
Other: Perspectives on pain — Understanding pain from a mind-body perspective and viewing pain as a stressor on physical sensations, thoughts, emotions, and behavior.
Other: Discussion — Discussion on patients' use of mindfulness to work with pain and pain-themed meditations.

SUMMARY:
This study will identify unique signatures that people have which can cause pain by evaluating biological, psychological, and social markers using artificial intelligence. These markers can be used to accurately predict the response of diverse individuals with chronic low back pain (cLBP) to Mindfulness-Based Stress Reduction. This will help enhance clinician decision-making and the targeted treatment of chronic pain.

The overall objective is to use a unique machine learning (ML) approach to determine the biomarker signature of persons undergoing mindfulness based stress reduction (MBSR) treatment for their chronic low back pain (cLBP). This signature will facilitate clinical prediction and monitoring of patient response to MBSR treatment.

The design of the study is a single-arm clinical trial of the evidence-based MBSR program for patients with cLBP.

DETAILED DESCRIPTION:
UG3 Phase Overview. The first 24-months of the project will be dedicated to performing machine learning modeling to identify candidate predictive and monitoring markers of cLBP response to MBSR, prior to the full clinical trial in the UH3 phase. We will also refine our procedures such as recruitment and outcomes assessment with 50 persons during the UG3 phase.

UH3 Phase Overview. Biopsychosocial markers will be identified of the response of diverse cLBP patients to MBSR (N=300) from comprehensive pain assessment and biopsychosocial data, including pain intensity and pain interference, physical activity, sleep, and heart rate for a 6-month period. Data will be collected and used for training and testing ML models. The MBSR program is evidence-based and meets weekly in a group via Zoom for 8-weeks for 90 minutes per week. Measures to determine biomarkers will be obtained at baseline (T1), four-weeks (T2), program completion (T3), four months (T4), and six months (T5). The main outcome timepoint with be at six months (T5), which allows time for durability of effects to be determined. The PEG (Pain, Enjoyment, General activity), obtained through online self-report surveys is the main outcome measure. Secondary outcomes of physical and psychological function will be self-report and obtained online, or if the patient prefers, by telephone, and physical activity, sleep, and heart rate variability will be collected by Fitbit.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain, which is pain that persists for at least 3-months and has resulted in pain on at least half the days in the past 6 months
* Willing and able to provide online or telephone informed consent
* Speak English as the intervention manual is currently written in English

Exclusion Criteria:

* Red flags- recent (past month) worsening of pain, unexplained fever, unexplained weight loss
* Pregnancy
* Metastatic cancer
* Not a patient at a participating clinic or persons not planning to continue as a patient at a participating clinic for 6 or more months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Pain, Enjoyment, General activity (PEG) composite score | 6 months
  The PEG is a 3-question scale: "pain average", "interference with general activity" and "interference with enjoyment of life". Each question is on a 0-10 scale, and total PEG is the average. Scores can range from 0-30 and <12=Mild,12 to <21 = Moderate, 21 to 30 = Severe chronic pain.

SECONDARY OUTCOMES:
Depression assessed by the eight-item Patient Health Questionnaire for Depression (PHQ-8) | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  The total score is determined by adding together the scores of each of the four items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
Anxiety assessed by the Generalized Anxiety Disorder-7 (GAD-7) | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Pain Self-Efficacy assessed by the Pain Self-Efficacy Questionnaire | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  The PSEQ is a 10-question survey that measures the confidence of a person with persistent pain to do a range of activities while in pain. The total score ranges from 0 to 60. High PSEQ scores are strongly associated with clinically- significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients. Higher scores (and a higher percentile) represent higher confidence to function with pain.
Catastrophizing assessed by the Pain Catastrophizing Scale Short Form | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  The Pain Catastrophizing Scale (PCS) measures three aspects of catastrophic cognitions about pain-rumination, magnification, and helplessness. It consists of 13 items scored from 0 to 4, with a total range of 0 to 52. Higher scores are less favorable and a score of more than 30 points may indicate clinical relevance.
Quality of Life assessed by the Patient Reported Outcomes Measurement Information System (PROMIS 29) | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  The PROMIS-29 v2. 0 profile measure assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items for each domain. HIgher scores indicate greater pain intensity.
Participants' Impression of change | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Patient Global Impression of Change (PGIC) will be used to assess this outcome. A score of 1=No change (or condition has got worse), 2 = Almost the same, hardly any change at all, 3 = A little better, but no noticeable change, 4 = Somewhat better, but the change has not made any real difference, 5 = Moderately better, and a slight but noticeable change, 6 = Better, and a definite improvement that has made a real and worthwhile difference 7 = A great deal better, and a considerable improvement that has made all the difference. A 2-point change is significant from the last reported score
Mindfulness assessed by the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  The CAMS-R is a 12-item measure designed to capture a broad conceptualization of mindfulness with language that is not specific to any particular type of meditation training. Items 2, 6, and 7 are reverse-scored. After appropriate reversals, values for items 1 - 12 are summed. Higher values reflect greater mindful qualities.
Sleep disturbance assessed by the PROMIS Sleep Disturbance-Short Form 6a | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  The PROMIS 6a scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days. The first two scale items assess sleep quality and the following 4 items assess domains of restfulness, sleep problems, and difficulty falling asleep. Each question has five response options ranging in value from one to five. To find the total raw score for a short so the range of scores is 6 to 30.
Pain-Sleep Duration | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  One question assesses sleep duration. This survey measures the impact of pain on the quality of sleep
Treatment components and effects assessed by the Healing Encounters and Attitudes List-Expectation | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Six questions ask about treatment expectancy. It assesses participants' attitudes towards and perceptions of treatment components that associated with nont specific treatment effects
Social support assessed by the Social Network Index | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  12 questions that ask about social support in regards to how many people a person sees and talk to regularly. The total score is calculated by finding the sum of the all items with a higher score indicating more social engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Morone, MD MS, Principal Investigator — Boston Medical Center; Jean King, PhD, Principal Investigator — Worcester Polytechnic Institute; Emmanuel Agu, PhD, Principal Investigator — Worcester Polytechnic Institute
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No